CLINICAL TRIAL: NCT04572451
Title: Phase I Study Investigating the Safety of Stereotactic Body Radiotherapy (SBRT) With Anti-PD1 and Anti-IL-8 for the Treatment of Multiple Metastases in Advanced Solid Tumors and Melanoma
Brief Title: Safety of SBRT With Anti-PD1 and Anti-IL-8 for the Treatment of Multiple Metastases in Advanced Solid Tumors and Melanoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yana Najjar (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Yana Najjar, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 20-228
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Melanoma; Unresectable Solid Tumors; Neoplasms; Neoplasms by Histologic Type; Neoplasms by Site; Antineoplastic Agents, Immunological; Antineoplastic Agents; Immune Checkpoint Inhibitors; Molecular Mechanisms of Pharmacological Action; Nivolumab
Keywords: Anti-PD-1 monoclonal antibody (mAb); Anti-IL-8; Stereotactic Body Radiotherapy (SBRT)
MeSH Terms: conditions — Melanoma; Neoplasms; Neoplasms by Histologic Type; Neoplasms by Site | interventions — Nivolumab; spartalizumab; HuMax-IL8; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nivolumab (Anti-PD-1) + BMS-986253 (Anti-IL-8) + SBRT (Experimental): 480 mg intravenous nivolumab (BMS-936558-01) every 4 weeks + 2,400 mg intravenous BMS-986253 (Anti-IL-8) every 2 weeks + Stereotactic Body Radiotherapy (SBRT)
  Interventions: Drug: nivolumab; Drug: BMS-986253; Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Drug: nivolumab — Nivolumab (BMS-936558-01), 480 mg intravenous (every 4 weeks)
  Treatment must be within 7 days of the last dose of radiation.
  Other Names: Opdivo®; Anti-PD-1
Drug: BMS-986253 — BMS-986253 (Anti-IL-8), 2,400 mg intravenous (every 2 weeks)
  Treatment must be within 7 days of the last dose of radiation.
  Other Names: Anti-IL-8
Radiation: Stereotactic Body Radiotherapy (SBRT) — Stereotactic Body Radiotherapy (SBRT) (varying doses)
  SBRT: Initial Dose fractionation of 3 or 5 fractions of radiation as determined by the location of the metastases to be irradiated, to at least 1 but no more than 4 metastatic lesions. There will be a minimum of 40 hours between treatments for an individual metastasis.
  SBRT must be completed within a 14-day window, separate from the screening phase. Treatment with nivolumab and BMS-986253 must be within 7 days of the last dose of radiation.

SUMMARY:
Nivolumab (and other agents affecting the anti-programmed death-1 [anti-PD-1] pathway) have demonstrated anti-tumor activity in multiple tumor types. Combinations of immune-oncology (IO) agents with complimentary mechanisms as well as radiation represent a promising strategy to improve response rates to immunotherapy and overcome resistance. In this phase I/Ib study, radiation will be used in combination with IO agents nivolumab and anti-IL-8 (BMS-986253) to assess toxicity by organ system and then assess the preliminary efficacy of the treatment regimen. In Part 1, the study will determine the safe doses of radiation by organ site in conjunction with nivolumab and BMS-986253. In Part 2, the treatment regimen will be investigated in melanoma, prioritizing acral melanoma, to describe the response rate to treatment as well as other clinical and safety outcomes. The study will also provide the opportunity to evaluate changes in the tumor microenvironment induced by the treatment.

DETAILED DESCRIPTION:
This is a study of SBRT in combination with nivolumab and BMS-986253, a monoclonal antibody (mAb) against human interleukin-8 (IL-8), conducted in humans with advanced solid tumors. This study will evaluate the safety profile, tolerability and preliminary efficacy of SBRT in combination with BMS-986253 and nivolumab in participants with advanced solid tumors and then specifically in melanoma, focused on acral melanoma. The study will be conducted in 2 parts.

Part 1 will evaluate the safety, tolerability of different doses of SBRT in combination with nivolumab (480 mg) and BMS-986253 (2400mg) every 2 weeks (Q2W) in participants with advanced solid tumors. This phase will begin with a cohort of participants who will receive a 2,400 mg flat dose of BMS-986253 Q2W combined with 480 mg flat dose of nivolumab Q4W along with SBRT (the dose is dependent on the irradiating organ).

Part 2 will assess preliminary efficacy of SBRT in combination with nivolumab and BMS-986253 in participants with advanced/metastatic/unresectable melanoma, focusing on acral melanoma, who progressed on anti-PD-(L)1 therapy.

This study aims to determine that safe doses will be found using ablative doses of SBRT with concurrent IO agents. Additional safety, tolerability and preliminary efficacy information in specific patient population will be gathered. Twenty participants with anti-PD-(L)1 refractory advanced/unresectable/metastatic melanoma, focusing on acral melanoma, will be enrolled into efficacy phase.

Note: The Sponsor-Investigator/Study Principal Investigator of this trial is Yana Najjar, MD at the University of Pittsburgh/UPMC. The Sponsor-Investigator of this trial at University of Chicago is Steven Chmura MD, PhD

ELIGIBILITY:
Inclusion Criteria:

* SAFETY COHORT

  1. Patients with advanced/metastatic/unresectable solid tumors progressed on standard therapies. Patients with melanoma and RCC will make up approximately 30% of total cohort.
  2. Patients with 1-4 tumor sites that can be irradiated safely
  3. Age > or equal 18 years
  4. ECOG performance status 0 or 1
  5. Patients must have normal organ and marrow function as defined below:

     * Leukocytes ≥ 3000/mcL;
     * absolute neutrophil count ≥ 1500/mcL;
     * Platelets ≥ 100,000/mcL;
     * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × upper limit of normal (ULN) ;
     * Total bilirubin ≤ 1.5 × ULN (except participants with Gilbert's Syndrome who must have normal direct bilirubin)
     * Serum creatinine ≤ 1.5 × ULN Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non- nodal lesions and short axis for nodal lesions) as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam
  6. Ability to understand and the willingness to sign a written informed consent document.
  7. Reproductive status

     * Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of study treatment.
     * Women must not be breastfeeding.
     * WOCBP must agree to follow instructions for method(s) of contraception (Appendix 5) for the duration of study treatment plus 5 half-lives of nivolumab plus 30 days (duration of ovulatory cycle), for a total of 155 days post treatment completion. Local laws and regulations may require use of alternative and/or additional contraception methods.
     * WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements, but should still undergo pregnancy testing as described in this section.
     * Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception (Appendix4) during combination treatment with study treatment BMS-986253 and nivolumab, plus 5 half-lives of nivolumab (∼125 days), plus 90 days (duration of sperm turnover), for a total of 215 days post-treatment completion. In addition, male participants must be willing to refrain from sperm donation during this time.
* EFFICACY COHORT

  1. Patients with anti-PD1/PDL1 refractory melanoma
  2. Patients with 1-4 tumor sites that can be irradiated safely
  3. Age ≥ 18 years
  4. ECOG performance status 0 or 1
  5. Patients must have normal organ and marrow function as defined above for safety cohort
  6. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non- nodal lesions and short axis for nodal lesions) as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam
  7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Known or suspected CNS metastases, with the following exceptions:

   a) Subjects with controlled brain metastases will be allowed to enroll. Controlled brain metastases are defined as no radiographic progression for at least 4 weeks following 18 radiation and/or surgical treatment at the time of randomization. b) Subjects must be off steroids for at least 2 weeks prior to initiation of investigational therapy c) Subjects with signs or symptoms of brain metastases are not eligible unless brain metastases are ruled out by computed tomography or magnetic resonance imaging.
2. Medical History and Concurrent Diseases

   * Patients who are receiving any other investigational agents.
   * History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab and BMS-986253
   * Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
   * Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

     i. Myocardial infarction (MI) or stroke/transient ischemic attack (TIA) within the 6 months prior to consent ii. Uncontrolled angina within the 3 months prior to consent iii. Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, torsades de pointes, or poorly controlled atrial fibrillation) within a month prior to consent iv. QTc prolongation > 480 msec v. History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, congestive heart failure with New York Heart Association [NYHA] functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, poorly controlled deep venous thrombosis, etc) vi. Cardiovascular disease-related requirement for daily supplemental oxygen vii. History of two or more coronary revascularization procedures within the 3 months prior to consent viii. Subjects with history of myocarditis, regardless of etiology
   * A confirmed history of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent
   * Subjects with history of life-threatening toxicity related to prior immune therapy (eg. anti-CTLA-4 or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) except those that are unlikely to re-occur with standard countermeasures (eg, hormone replacement after endocrinopathy).
   * Subject has been administered prior chemotherapy or immunotherapy at any time, and any with radiation therapy within 4 weeks prior to time of consent or who has not recovered (ie, ≤ Grade 1 or at baseline) from adverse events due to previously administered agent.

     1. Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
     2. Subjects with endocrinopathy which is adequately controlled with hormone replacement therapy are an exception to this criterion and may qualify for the study.
   * If subject underwent major surgery, subject must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
   * Subject has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
   * A known or underlying medical condition that, in the opinion of the investigator could make the administration of study drug hazardous to the subject or could adversely affect the ability of the subject to comply with or tolerate study therapy.
   * Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated with the study drugs.
   * Subjects who are unable to undergo venipuncture and/or tolerate venous access
   * Evidence of active infection that requires systemic antibacterial, antiviral, or antifungal therapy ≤ 7 days prior to initiation of study drug therapy
   * Subjects who are on immunosuppressive therapy (systemic steroids 10mg and more daily use)
   * Prisoners or subjects who are involuntarily incarcerated
   * Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness
   * Inability to comply with restrictions and prohibited activities and treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Dose Limiting Toxicities (DLT) | Up to 8 weeks after start of immunotherapeutic treatment
  The rate of Dose Limiting Toxicities (DLT) that are determined to be definitely, probably or possibly attributed to SBRT or one or both of the immunotherapies. Patients receiving one of more fractions of SBRT are evaluable for DLT. Toxicities include grade 3 or higher adverse events, by organ system, by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Incidence of grade 3 or higher adverse events | Up to 1 year after start of immunotherapeutic treatment
  Incidence of grade 3 or higher adverse events, by organ system, per CTCAEv5.0, determined to be definitely, probably or possibly attributed to SBRT or one or both of the immunotherapies.
Objective Response | Up to 3 years
  The proportion of patients that experience a Complete Response (CR) or Partial Response (PR) per RECIST v1.1. Per RECIST v1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Progression-free survival (PFS) | Up to 3 years
  The duration of time from first day of treatment until disease progression or date of death from any cause will be estimated with a 90% confidence interval. Progression as defined by RECIST v1.1 for target lesions: Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions: Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Overall survival (OS) | Up to 3 years
  Overall survival (OS) (of the cohort) which is defined as elapsed time from date of first treatment until date of death.
Local tumor control (RECIST v1.1) | Up to 3 years
  The total disappearance of the primary tumor and neighboring lymph node metastases without any local recurrence on long-term follow-up, per RECIST version 1.1. Complete response per RECIST v1.1 is the disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm.
Local tumor control (irRECIST) | Up to 3 years
  The total disappearance of the primary tumor and neighboring lymph node metastases without any local recurrence on long-term follow-up, by immune-related RECIST (irRECIST). Immune Complete Response (iCR) is the complete resolution of non-nodal lesions and < 10 mm short-axis for lymph nodes. No confirmation necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Yana Najjar, MD, FACP, Principal Investigator — UPMC Hillman Cancer Center
Locations (2):
- United States (2):
  - University of Chicago Medical Center, Chicago, Illinois
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No